CLINICAL TRIAL: NCT04455152
Title: Self-control Intervention to Increase Adherence to Web-based Self-help for Body-focused Repetitive Behaviors
Brief Title: Self-control and Body-focused Repetitive Behaviors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: American University (Other)
Responsible Party: Principal Investigator, David A. F. Haaga, Professor of Psychology, American University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Mellon2020CAS
Record Dates: First submitted 2020-06-29; First posted 2020-07-02 (Actual); Last update posted 2022-11-07 (Actual); Status verified 2022-11

CONDITIONS: Trichotillomania (Hair-Pulling Disorder); Skin-Picking
MeSH Terms: conditions — Trichotillomania; Excoriation Disorder

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to self-control vs. wait list for 2 weeks after baseline assessment and before all receive 10 weeks of web-based self-help.
Who Masked: Investigator
Masking Description: Random assignment will not be made, nor known to anyone, until informed consent process and baseline assessment are completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-control (Experimental): two-week period of practicing self-control (attempting to avoid eating sweet foods) and self-monitoring success in doing so
  Interventions: Behavioral: self-control
- wait list (No Intervention): waiting 2 weeks after baseline assessment before gaining access to web-based self-help

INTERVENTIONS:
Behavioral: self-control — avoiding eating sweets as a way of building self-control strength
  Arms: Self-control

SUMMARY:
Web-based self-help could work well to disseminate behavior therapies for body-focused repetitive behaviors (BFRB) such as hair pulling and skin picking. Previous research suggests that this method works well for people who use the program a great deal, but many participants do not. Adhering frequently to a BFRB self-help program requires self-control because the costs occur immediately (time, trouble, possible boredom), whereas the benefits (reduced symptoms) are realized later.

This study will test whether two weeks of practice of a self-control exercise (avoiding consumption of sweet foods), compared to wait list, will increase adherence during a subsequent 10-week trial of BFRB self-help.

DETAILED DESCRIPTION:
Body-focused repetitive behaviors (BFRB) such as hair pulling and skin picking are prevalent and associated with distress and impairment. Behavioral treatments of BFRB are effective, but access to therapists with expertise in them is limited. One way to reduce the access problem is to disseminate evidence-based treatments in the form of web-based self-help programs. Behavior therapy methods are incorporated in such programs for hair pulling and skin picking, each of which appears promising based on uncontrolled studies. The investigators conducted the first randomized controlled trial of stop pulling.com. Compared to wait list, those with access to the program showed a small but significant advantage in reduction of interviewer-rated TTM symptoms. However, there was no significant difference from wait list on self-reported symptoms, alopecia [hair loss severity], impairment, or quality of life.

Average outcomes of stop pulling.com were thus modest, but the investigators see a couple of ways to extend this work in the proposed project. First, the coverage of BFRB is expanded by including stop picking.com. Second, web-based self-help will be tested as a free-standing intervention, the way it is offered to the public. In the previous research, stop pulling.com was the first phase of a stepped care program, to be followed [if desired] by in-person therapy. This could have biased the sample by limiting it to residents of the Washington, DC area and by attracting some who were not interested in web-based self-help and only wanted the in-person therapy. Consistent with this concern, 19% of participants never tried the self-help program. Third and most importantly, a preliminary self-control intervention intended to increase adherence to web-based self-help will be tested. Nonadherence is the main problem for self-help in behavioral health in general, and in BFRB in particular. In the earllier study of stop pulling.com, participants logged on and entered data on a median of just 12.5 days (out of the intended 70) in a 10-week span. Those who used it more tended to get more benefit, but the challenge is how to increase adherence overall.

Adherence to web-based self-help may be seen as requiring self-control because its costs are borne immediately (e.g., somewhat tedious assessments such as self-monitoring logs), whereas the benefits are probabilistic and delayed (reduction of symptoms over a period of weeks). Just as someone taking up a new exercise routine has to do something effortful and perhaps disagreeable at first in order to (likely) gain later benefits, so too the person with a BFRB needs to log data regarding urges or pulling/picking episodes in a meticulous manner in the hope of eventually getting useful individualized suggestions, implementing them, and (probably) reducing symptom severity. The method for improving self-control to be tested in this project derives from the "strength" model of self-control, in which willpower is considered analogous to a muscle. Research supports two key implications of this model, that exertion of self-control temporarily depletes capacity and impairs performance on other tasks (e.g., holding a hand grip as long as one can makes it harder to choose a healthy snack rather than chocolate), but that practicing self-control builds up self-control strength over time.

Approach: In this study 40 participants (20 hair pullers, 20 skin pickers-10 of each in each experimental condition) will be randomly assigned after a pretest of BFRB severity to one of two conditions: (a) 2-week self-control task vs. (b) 2-week wait list, followed in each condition by paid access to web-based self-help for 10 weeks and then post-test. The self-control intervention asks the participant to avoid eating sweet foods and to report via email each day how well they were able to do so. Smokers who performed this task were significantly better able to maintain abstinence after smoking cessation than were those in a control condition. The main dependent variable will be adherence, the number of days (out of 70) on which the participant logged in and entered data on their behavior. Secondary outcomes include change in BFRB symptoms and qualitative feedback on the self-control task and the self-help program.

ELIGIBILITY:
Inclusion Criteria:

* meet the diagnostic criteria for either Hair Pulling Disorder (trichotillomania) or Skin Picking Disorder
* have regular access to the Internet
* age 18 or older

Exclusion Criteria:

[all current, not lifetime]

* suicidal thoughts
* major depression
* psychosis
* severe anxiety
* substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

PRIMARY OUTCOMES:
Adherence | 10 weeks
  number of days (of maximum 70) on which participant logged into self-help program and entered data

SECONDARY OUTCOMES:
BFRB symptoms | 12 weeks
  depending on participant's primary problem, either hairpulling or skin picking severity
program feedback | week 12 only
  qualitative feedback on self-control task and on web-based self-help

CONTACTS AND LOCATIONS:
Locations (1):
- American University, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data could be shared with other researchers
Supporting Information: Study Protocol, SAP, ICF
Time Frame: a year after completion of data collection, available indefinitely
Access Criteria: Any faculty member, or graduate student collaborating with a faculty member.